CLINICAL TRIAL: NCT03250416
Title: The First Affiliated Hospital of Chongqing Medical University
Brief Title: Management of Noninvasive Ventilation in Hypoxemic Patients
Status: Completed | Type: Observational
Sponsor: Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Duan jun, Doctor, Chongqing Medical University
Other Study IDs: ChongqingMU2
Record Dates: First submitted 2017-08-11; First posted 2017-08-15 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Noninvasive Ventilation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigator aimed to manage noninvasive ventilation in patients with hypoxemic respiratory failure.

DETAILED DESCRIPTION:
Patients with hypoxemic respiratory failure were enrolled in this study. The investigator collected the data at beginning and first stage of noninvasive ventilation to analyze the efficacy of noninvasive ventilation. To manage the noninvasive ventilation easily, the investigator also aimed to develop a scale to predict the efficacy of noninvasive ventilation, and used this scale to guide clinicians how to use noninvasive ventilation.

ELIGIBILITY:
Inclusion Criteria:

* PaO2/FiO2 less than 300; PaCO2 less than 50 mmHg; Respiratory rate more than 25 breaths/min or presence of labored breath.

Exclusion Criteria:

* Requirement of emergency intubation; Sequential use of noninvasive ventilation after extubation;Use of noninvasive ventilation after accident extubation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The main population is acute hypoxemic respiratory failure. The subgroup included ARDS, pneumonia, sepsis and so on.
Sampling Method: Non-Probability Sample
Enrollment: 2179 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Noninvasive ventilation failure | From participation to 30 days
  Noninvasive ventilation failure was defined as requirement of intubation.

SECONDARY OUTCOMES:
Mortality | From participation to 30 days
  Mortality in ICU and hospital
ICU stay | From participation to 30 days
  Length of ICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Jun Duan, Dr, Principal Investigator — First Affiliated Hospital of Chongqing Medical University
Locations (1):
- The First Affiliated Hospital ,Chongqing Medical Univercity, Chongqing, Chongqing Municipality, China